CLINICAL TRIAL: NCT02219633
Title: An Explorative Trial Evaluating the Effect of LEO 39652 Cream in Adults With Mild to Moderate Atopic Dermatitis (AD)
Brief Title: Effect of LEO 39652 Cream in Adults With Mild to Moderate Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0083-1085; 2014-000849-80 (EudraCT Number)
Record Dates: First submitted 2014-08-13; First posted 2014-08-19 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2016-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 39652 cream (Experimental): Topical application
  Interventions: Drug: LEO 39652 cream
- LEO 39652 cream vehicle (Placebo Comparator): Topical application
  Interventions: Drug: LEO 39652 cream

INTERVENTIONS:
Drug: LEO 39652 cream — Applied for 21 days

SUMMARY:
The aim of this trial is to assess the efficacy of LEO 39652 cream compared with LEO 39652 cream vehicle in adults with mild to moderate AD after 3 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Atopic Dermatitis (AD) as defined by Hanifin and Rajka criteria and with mild to moderate disease severity (IGA 2 or 3)
* Two symmetrical and comparable Entire Treatment Areas, on the same body region (left and right part)
* Subjects must be in good health
* Female subjects of childbearing potential and male subjects must be willing to consent to using high effective methods of contraception

Exclusion Criteria:

* Any condition in the treatment areas that in the opinion of the investigator could interfere with clinical assessments, e.g. acne, infection, rash (other than atopic dermatitis), sunburn, hyper-or hypopigmentation, scars
* Dark-skinned persons (i.e. skin type IV to VI according to Fitzpatrick classification system) whose skin colour prevents reliable clinical assessments
* Any permanent (or transient within 28 days prior to dosing) disease (in particular cardiac disease such as heart failure or history of myocardial infarction) that may interfere with the subjects safe participation in the trial, with the subjects ability to participate in the trial or with the clinical assessments
* Subjects with congenital or acquired immunodeficiencies or in subjects on therapy that causes immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Total sign score at end of treatment | 22 days
  Total Sign Score is defined as the sum of severity scores (4-point scale) of the Individual Sign Scores(erythema, edema/papulation, oozing/crusting, excoriations, lichenification and dryness)for each assessed area.

SECONDARY OUTCOMES:
Total sign score on limited treatment area | 22 days
Investigator's treatment area assessment of disease severity | 22 days
Subject´s treatment area assessment of disease severity | 22 days
Subject´s assessment of itching | 22 days
Transepidermal Water Loss | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Graßhoff, MD, Principal Investigator — Proinnovera GmbH
Locations (1):
- proinnovera GmbH, Center of Dermatology Excellence, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en